CLINICAL TRIAL: NCT02483169
Title: Double Blind Placebo Controlled Multicenter Trial for Prevention of IMT Progression in the Ischemic Stroke Patients With High Risk of Cerebral Hemorrhage With Cilostazol and Probucol
Brief Title: PreventIon of IMT Progression in iSchemic Stroke Patients With High Risk of Cerebral HemOrrhage-IMT Study
Acronym: PICASSO-IMT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Sun U. Kwon, Professor, Asan Medical Center
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PICASSO-IMT
Record Dates: First submitted 2015-06-24; First posted 2015-06-26 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Brain Ischemia; Intracranial Hemorrhages
Keywords: ischemic stroke; intracranial hemorrhage; cilostazol; probucol; intima media thickness
MeSH Terms: conditions — Brain Ischemia; Intracranial Hemorrhages; Ischemic Stroke | interventions — Cilostazol; Probucol; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cilostazol+ Probucol (Experimental): 100mg cilostazol bid plus probucol plus placebo of aspirin
  Interventions: Drug: cilostazol; Drug: Probucol; Drug: Placebo of aspirin; Device: Intima-medial thickness
- Aspirin + Probucol (Active Comparator): aspirin plus placebo cilostazol plus probucol
  Interventions: Drug: Probucol; Drug: Aspirin; Drug: placebo of cilostazol; Device: Intima-medial thickness
- Cilostazol (Experimental): cilostazol plus placebo of aspirin
  Interventions: Drug: cilostazol; Drug: Placebo of aspirin; Device: Intima-medial thickness
- Aspirin (Active Comparator): aspirin plus placebo of cilostazol
  Interventions: Drug: Aspirin; Drug: placebo of cilostazol; Device: Intima-medial thickness

INTERVENTIONS:
Drug: cilostazol — Cilostazol 100mg bid
  Other Names: Pletaal produced by Korea Otsuka Pharmaceutical company
  Arms: Cilostazol; Cilostazol+ Probucol
Drug: Probucol — Probucol 250mg bid
  Other Names: Probucol is produced by Otsuka Pharmaceutical
  Arms: Aspirin + Probucol; Cilostazol+ Probucol
Drug: Aspirin — Aspirin 100mg qd
  Arms: Aspirin; Aspirin + Probucol
Drug: placebo of cilostazol — same shape and size of active cilostazol
  Arms: Aspirin; Aspirin + Probucol
Drug: Placebo of aspirin — same size and shape of active aspirin 100mg
  Arms: Cilostazol; Cilostazol+ Probucol
Device: Intima-medial thickness — ultrasound measured IMT of both common carotid arteries
  Other Names: - Annualized change of mean and maximum common carotid intima-medial thickness; - Annualized change of carotid plaque score

SUMMARY:
Through this study, the investigators are to prove that Cilostazol effectively prevent progression of intima-medial thickness in ischemic stroke patients with high risk of cerebral hemorrhage, along with no significant increase in the risk of occurrence of hemorrhagic side effects.

The primary hypothesis of this study is; Cilostazol alone or with probucol will reduce the progression of intima-medial thickness compared to aspirin in the ischemic stroke patients with symptomatic or asymptomatic old cerebral hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ischemic stroke within 120 days
* Adult aged 20 years or older
* High risk of hemorrhagic stroke (history of intracranial hemorrhage or imaging evidence of previous intracranial hemorrhage)
* Informed consent

Exclusion Criteria:

* Clinical diagnosis of myocardial infarction or coronary intervention within 4 weeks
* Bleeding tendency
* Pregnant or breast-feeding woman
* Hemorrhagic stroke within 6 months
* Patient who was taking antithrombotic medication other than aspirin and does not agree to change the previous medication
* Severe cardiovascular disease such as cardiomyopathy or congestive heart failure
* Life expectancy less than one year
* Contraindication to long term aspirin use
* Enrolled in other clinical trial within 30 days

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2009-06; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
mean carotid IMT progression | one year
  Annualized rate of change in mean common carotid intimal-medial thickness

SECONDARY OUTCOMES:
maximum carotid IMT progression | one year
  annualized rate of change in maximal carotid intimal-medial thickness
carotid plaque score | one year
  annualized change of carotid plaque score

CONTACTS AND LOCATIONS:
Overall Officials: Sun U Kwon, MD,PhD, Principal Investigator — Department of Neurology, Asan Medical Center